CLINICAL TRIAL: NCT06964022
Title: Impact of Blood-Flow-Restriction Prehabilitation on Pre- and Postoperative Rehabilitation After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023_D
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis (OA) of the Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Control (Active Comparator): Participants of this group were active controls, exercising with a sham-BFR intervention during prehabilitation.
  Interventions: Other: Sham-BFR
- Intervention Group (Experimental): Participants of this group were exercising with a BFR intervention during prehabilitation.
  Interventions: Other: BFR

INTERVENTIONS:
Other: Sham-BFR — Six-week prehabilitation program (2/week): Unilateral Leg Press and Leg extension exercise with 30% of the individual 1RM by using a sham-BFR intervention with 20mmHg exercise pressure.
  Arms: Active Control
Other: BFR — Six-week prehabilitation program (2/week): Unilateral Leg Press and Leg extension exercise with 30% of the individual 1RM by using a BFR intervention with an exercise pressure corresponding to 60% of the individual LOP.
  Arms: Intervention Group

SUMMARY:
Degenerative and traumatic diseases of the musculoskeletal system lead to increased immobility of a patient, which in turn results in muscle atrophy. BFR training is a training method in which a blood pressure cuff partially blocks the arterial blood flow to the exercising limb and completely blocks the venous blood flow. During exercise, an externally induced venous occlusion occurs. This stimulus increases the metabolic stimulus in the occluded extremity - this means that strength can be increased even with low weights, which is why this training is also suitable for people who should not use high training loads due to injuries or operations.

ELIGIBILITY:
Inclusion Criteria:

* Indication for TKA Surgery
* Ability to perform prehabilitation exercise

Exclusion Criteria:

* Sickle Cell Anemia
* Iatrogenic changes in the vessels of the lower extremities (e.g. stents)
* Open wounds/Infection of the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Subjective Pain Value | Pre- to 6 weeks Post Surgery
  Subjective pain perception, assessed by visual analog scale (0-100mm)
Muscle Strength | Pre- to 6 weeks Post Surgery
  Muscle Strength assessed by isometric maximal test (Nm)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No